CLINICAL TRIAL: NCT02554539
Title: Human Embryonic Transciptomic Modification Induced by miRNAs Secreted by Human Endometrium to Endometrial Fluid
Brief Title: Transciptomic Modification Induced by miRNAs in Endometrial Fluid
Acronym: miRNA_EF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Meera Sridhar Shah, Clinical Fellow, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 34225
Record Dates: First submitted 2015-08-27; First posted 2015-09-18 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: MicroRNA in Endometrial Fluid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Obese (Experimental): Women, aged 21-45 with BMI >30
  Interventions: Procedure: Endometrial fluid aspiration
- Normal weight (Experimental): Women, aged 21-45 with BMI < 25
  Interventions: Procedure: Endometrial fluid aspiration

INTERVENTIONS:
Procedure: Endometrial fluid aspiration — Patient will undergo a biopsy to aspirate endometrial fluid from the uterine cavity

SUMMARY:
The purpose of this study is to understand the mechanism of communication between the uterine environment and the preimplantation human embryo. The investigators are interested in understanding how the in-utero environment during the window of implantation is different in normal weight and overweight/obese women and how this may impact the programming of the developing embryo.

ELIGIBILITY:
Inclusion Criteria:

* Meet the WHO criteria for normal weight (BMI < 25) and overweight/obese (BMI > 25)
* Age 21-45

Exclusion Criteria:

* Age < 21 or > 45
* Women with history of hysterectomy

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Gene expression profile in human embryos | Samples will be collected within 1 month of enrollment
  We will perform RNA sequencing on the human embryo to quantify which genes are up and down regulated in obese compared to normal weight controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States